CLINICAL TRIAL: NCT01077453
Title: Phase I Dose-Finding Trial of Letrozole in Postmenopausal Women at High Risk for Breast Cancer
Brief Title: Letrozole in Preventing Breast Cancer in Healthy Postmenopausal Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2013-00757; NCI-2013-00757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-0869-04 (Other: University of Arizona Health Sciences Center); UAZ08-12-02 (Other: DCP); N01CN35158 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy, no Evidence of Disease; Lobular Breast Carcinoma in Situ
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Arm I (2.5 mg letrozole) (Experimental): Patients receive 2.5 mg of letrozole PO thrice weekly for 6 months.
  Interventions: Drug: letrozole; Other: quality-of-life assessment; Other: laboratory biomarker analysis
- Arm II (1.0 mg letrozole) (Experimental): Patients receive 1.0 mg of letrozole PO thrice weekly for 6 months.
  Interventions: Drug: letrozole; Other: quality-of-life assessment; Other: laboratory biomarker analysis
- Arm III (0.25 mg letrozole) (Experimental): Patients receive 0.25 mg of letrozole PO thrice weekly for 6 months.
  Interventions: Drug: letrozole; Other: quality-of-life assessment; Other: laboratory biomarker analysis
- Arm IV (2.5 mg letrozole) (Experimental): Patients receive 2.5 mg of letrozole PO once daily for 6 months.
  Interventions: Drug: letrozole; Other: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: letrozole — Given orally
  Other Names: CGS 20267; Femara; LTZ
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects and the best dose of letrozole in preventing breast cancer in healthy postmenopausal women at high risk for breast cancer. Chemoprevention is the use of drugs to keep breast cancer from forming or coming back. The use of letrozole may keep cancer from forming in healthy postmenopausal women at high risk for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the effect of lower and intermittent doses of letrozole to standard letrozole therapy on estrogen suppression in postmenopausal women at high risk for developing breast cancer.

SECONDARY OBJECTIVES:

I. Comparison of the effect of lower and intermittent doses of letrozole to standard therapy on signs and symptoms of estrogen deficiency, including menopausal symptoms, serum lipid profile, and serum marker of bone turnover.

II. Comparison of the effect of lower and intermittent doses of letrozole to standard therapy on nuclear chromatin abnormality of breast epithelial cells collected by random periareolar fine needle aspiration (RPFNA).

TERTIARY OBJECTIVES:

I. Determine the prevalence of breast cancer stem cells in the fine needle breast aspirates and explore the potential intervention effect on the prevalence of breast cancer stem cells.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive 2.5 mg of letrozole orally (PO) thrice weekly for 6 months.

ARM II: Patients receive 1.0 mg of letrozole PO thrice weekly for 6 months.

ARM III: Patients receive 0.25 mg of letrozole PO thrice weekly for 6 months.

ARM IV: Patients receive 2.5 mg of letrozole PO once daily for 6 months.

After completion of study treatment, patients are followed up at week 30.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women at "high risk" for breast cancer will be eligible for the study; definition of menopause will be:

  * Amenorrhea for at least 12 months, or
  * History of hysterectomy and bilateral salpingo-oophorectomy, or
  * At least 55 years of age with prior hysterectomy with or without oophorectomy, or
  * Age 35 to 54 with a prior hysterectomy without oophorectomy OR with a status of ovaries unknown with documented follicle-stimulating hormone level demonstrating elevation in postmenopausal range
  * "High risk" for breast cancer will be defined as:

    * Prior histologically confirmed lobular carcinoma in situ (LCIS) treated by local excision only, or
    * At least 1.66% probability of invasive breast cancer within 5 years using the Breast Cancer Risk Assessment Tool
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1; Karnofsky 80% or above
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 X institutional ULN
* Creatinine =< 1 X institutional ULN
* Recent mammogram negative for breast cancer, Breast Imaging-Reporting and Data System (BIRADS) score < 3 (within the last 12 months)
* Ability to understand and the willingness to sign a written informed consent document; only potential participants with the ability to understand and the willingness to sign a written document will be presented with an informed consenting document

Exclusion Criteria:

* Women diagnosed with osteoporosis (previously or on screening dual-energy X-ray absorptiometry [DEXA] for this study) and not on a stable dose of long or short-acting bisphosphonates therapy for at least 3 months will be excluded from the study; women diagnosed with osteoporosis and on raloxifene (Evista) therapy will be excluded from the study; use of calcium and/or vitamin D for osteoporosis prevention or treatment is allowed; women with osteopenia will be allowed to participate in this study
* Have had invasive cancer within the past five years except non-melanoma skin cancer
* Evidence of suspicious of malignant disease on bilateral mammogram within the past year unless ruled out by further evaluation
* History of prior invasive breast cancer or intraductal carcinoma in situ, or history of prior radiation therapy to the chest or breast
* Participants may not be receiving any other investigational agents; participants may not be concurrently enrolled in another breast cancer prevention intervention trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to letrozole
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Within 3 months since prior estrogen or progesterone replacement therapy, oral contraceptives, androgens, luteinizing hormone-releasing hormone analogs, prolactin inhibitors, or antiandrogens
* Within 3 months since prior tamoxifen, raloxifene, or other selective estrogen-receptor modulators
* Within 3 months since regular use (more than 2 times a week) of prior estrogenic supplements or herbal remedies
* History of bleeding or clotting disorder; current or recent (within 3 months) use of Coumadin, Plavix or other systemic anticoagulant other than aspirin is not permitted if subject chooses to participate in the optional RPFNA procedure; if a subject chooses not to participate in the RPFNA procedure, prior or current treatment with systemic anticoagulants is permitted

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percentage of serum estradiol suppression in postmenopausal women at high risk for breast cancer | Baseline to week 30
  Three one-sided two-sample t-tests will be conducted on the ratios of the mean percentage of suppression simultaneously to test for non-inferiority. A multivariate t-distribution is used to derive the critical value and the power.

SECONDARY OUTCOMES:
Change in serum estrone levels | Baseline to week 30
  Three one-sided two-sample t-tests will be performed to evaluate the ratio of the mean changes (or percentage of changes) of each of the three intermittent dosing groups to that of the standard therapy control group simultaneously for each of the endpoints at an overall significance level of 5%.
Change in serum testosterone levels | Baseline to week 30
  Three one-sided two-sample t-tests will be performed to evaluate the ratio of the mean changes (or percentage of changes) of each of the three intermittent dosing groups to that of the standard therapy control group simultaneously for each of the endpoints at an overall significance level of 5%.
Menopausal symptoms as assessed by quality of life measures, as assessed by Medical Outcomes Study 36-item Short Form Health Survey (SF-36) and Menopause Specific Quality of Life Questionnaire (MENQOL) | Up to week 30
Nuclear chromatin abnormality as assessed by karyometry | Up to week 30

OTHER OUTCOMES:
Prevalence of breast cancer stem cells by the proportion of aldehyde dehydrogenase positive cells, assessed by the Aldeflour assay | Up to week 30
Relative expression of stem cell markers to housekeeping genes, assessed by quantitative real time polymerase chain reaction | Up to week 30

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lopez, Principal Investigator — University of Arizona Health Sciences Center
Locations (3):
- United States (3):
  - Arizona Cancer Center - Tucson, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Lopez AM, Pruthi S, Boughey JC, Perloff M, Hsu CH, Lang JE, Ley M, Frank D, Taverna JA, Chow HH. Double-Blind, Randomized Trial of Alternative Letrozole Dosing Regimens in Postmenopausal Women with Increased Breast Cancer Risk. Cancer Prev Res (Phila). 2016 Feb;9(2):142-8. doi: 10.1158/1940-6207.CAPR-15-0322. Epub 2015 Dec 14. PMID 26667449